CLINICAL TRIAL: NCT02819713
Title: Difference in Pain Perception by Patients With Prostate Biopsy Using Instillagel Compared Guided Ultrasound Gel, a Randomized Controlled Trial
Brief Title: Difference in Pain Perception by Patients With Prostate Biopsy Using Instillagel Compared With Guided Ultrasound Gel
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: LTC-744-040111-Roelofs; NL35454.091.11 (Other: CMO regio Arnhem-Nijmegen)
Record Dates: First submitted 2011-08-08; First posted 2016-06-30 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Prostate Biopsy
Keywords: Prostate Biopsy; NRS-score; instillagel; ultrasound conductive gel
MeSH Terms: interventions — chlorhexidine gluconate, lidocaine drug combination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ultrasound gel (Placebo Comparator)
  Interventions: Other: ultrasound gel
- Instillagel (Active Comparator)
  Interventions: Other: Instillagel

INTERVENTIONS:
Other: ultrasound gel
  Arms: ultrasound gel
Other: Instillagel
  Arms: Instillagel

SUMMARY:
This is a randomized controlled trial. One group (intervention group) will get in advance to the prostate biopsy rectal approximately 5 cc Instillagel. And one group (control group) will get in advance to the ultrasound -guided prostate biopsy rectal gel. Pain is measured using the Numerical Rating Scale (NRS). The NRS is an imaginary line from 0 until 10. The 0 is no pain and 10 is most worst imaginable pain.

DETAILED DESCRIPTION:
Urologist within Rijnstate use both Instillagel and ultrasound gel during prostate biopsy. According to the protocol, the ultrasound-guided prostate biopsy must be performed using ultrasound gel. Some urologists departed from the protocols because they think that Instillagel will give a pain reduction. With this research we investigate whether Instillagel will have an effect on the pain perception bij the patients.

There will be three moments of pain measurements; Prior to het prostate biopsy. Immediately after the prostate biopsy. And five to thirty minutes after the prostate biopsy, when the patient is dressed and before the patient goes home.

Primary endpoint Pain measured by the Numeric Rating Scale

Secondary endpoints

* Age of patient
* Previous prostate biopsy
* The number of biopsies taken
* Presence of prostate cancer
* Other complications as after prostate biopsy

The prostate biopsy will be performed by a urologist working at the outpatient clinic of Rijnstate. The ultrasound equipment that will be used during prostate biopsy is Aloka ProSound SSD-3500 or Aloka ProSound SSD or SV-3500 SX.

ELIGIBILITY:
Inclusion Criteria:

* outpatient ultrasound guide prostate biopsy
* > 40 years old.
* Good knowledge of dutch language

Exclusion Criteria:

* coagulation disorders
* disorders of the rectum like hemorrhoids, anal fistula, proctitis, rectal polyps and rectal cancer.
* treated for active urinary tract infection
* known of allergy to lidocaine
* taking antidepressants
* using anaesthetic agents
* neurological disorders such as Parkinsons disease, hernias and spinal cord injury
* treated with radiotherapy for prostate cancer

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
NRS score | Three measurements before, just after and 5 -30 minutes after procedure

SECONDARY OUTCOMES:
age of patient | Two weeks after the prostate biopsy.
Previous prostate biopsy | Two weeks after the prostate biopsy.
The number of biopsies taken | two weeks after prostate biopsy
Other complications as after prostate biopsy | two weeks after prostate biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Marita van den Berg, Principal Investigator — Rijnstate Hospital
Locations (1):
- Rijnstate location Arnhem, Arnhem, Gelderland, Netherlands